CLINICAL TRIAL: NCT01832558
Title: The EPOCH Study (Eplerenone on Top of ACE Inhibition in Chronic Kidney Disease Patients With Hypertension)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marcus Saemann, Assoc. Prof. Priv.-Doz. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT: 2012-002175-34
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: CKD II-III
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Eplerenone (Experimental): Eplerenone 25-50mg daily additionally to standard ACE-inhibition with enalapril 20mg daily
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator): Placebo additionally to standard ACE-inhibition with enalapril 20mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone
  Arms: Eplerenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
In a prospective single centre placebo-controlled trial over ten weeks, 24 CKD II-III patients (eGFR 30-89 ml/min per 1.73 m2) with DM II will be randomized to enalapril 20mg per day after a two week run-in phase. Thereafter, patients will either receive eplerenone 25mg (n=12) or a placebo (n=12) for eight weeks. Eplerenone will be increased to 50mg under close monitoring of serum potassium levels. Employing a novel mass-spectrometry ( MS)-based method, quantification of up to 10 different Ang metabolites (Ang I, Ang II, Ang 1-7, Ang 1-9, Ang 2-10, Ang 1-5, Ang 2-7, Ang 3-7, Ang 3-8 and Ang 2-8) will be performed simultaneously out of blood sera (after run-in phase and after 10 weeks).

ELIGIBILITY:
Inclusion Criteria:

* CKD II to III and diabetes mellitus type 2
* CKD will be defined according to estimated glomerular filtration rate (eGFR) with the MDRD formula
* eGFR between 30 and 89 ml/min
* albumin excretion rates > 300 mg/24 hours (UACR > 300 mg/gram) or > 200 mg/g if already receiving any RAS blockade Patients should be hypertonic stage I or II according to the European guidelines (Chobanian et al. JAMA 2003)

Exclusion Criteria:

* Age < 18 years
* UACR > 3500mg/g
* severe hypertension
* pregnancy
* unwilling or inability to sign the informed consent
* coronary heart disease
* systolic blood pressure < 130 mmHg
* additional RAS interfering drugs (ACEis, ARBs, direct renin inhibitors)
* 25-hydroxy vitamin D levels below 16.6±8.3 pg/ml
* 1,25-dihydroxy vitamin D 33.1±15.5 pg/ml

Intolerance to eplerenon or an excipient of it:

tablettcore: Lactose-Monohydrat Mikrokristalline Cellulose (E 460) Croscarmellose-sodium (E 468) Hypromellose (E 464) Sodiumdodecylsulfat Talkum (E 553b) Magnesiumstearat (E 470b)

filmcoat

Opadry, yellow:

Hypromellose (E 464) Titandioxid (E 171) Macrogol 400 Polysorbat 80 (E 433) Yellow ironoxide (E 172) Red ironoxide (E 172)

* Patients with Serumpotassium > 5,0 mmol/l at start of the treatment
* Patients with severe renal insufficiency (eGFR <30ml/min./1.73 m2)
* Patients with severe liver insufficiency (Child-Pugh class C)
* Patients taking potassium saving diuretics, potassium supplements or strong CYP3A4-inhibitors (z. B. Itraconazol, Ketoconazol, Ritonavir, Nelfinavir, Clarithromycin, Telithromycin und Nefazodon)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-11; Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Angiotensin levels (pg/ml) of CKD II-III patients with DM II with eplerenone additional to enalapril in comparison to patients who receive a placebo on top of enalapril therapy. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Shavit L, Lifschitz MD, Epstein M. Aldosterone blockade and the mineralocorticoid receptor in the management of chronic kidney disease: current concepts and emerging treatment paradigms. Kidney Int. 2012 May;81(10):955-968. doi: 10.1038/ki.2011.505. Epub 2012 Feb 15. PMID 22336987
- [Background] Epstein M, Williams GH, Weinberger M, Lewin A, Krause S, Mukherjee R, Patni R, Beckerman B. Selective aldosterone blockade with eplerenone reduces albuminuria in patients with type 2 diabetes. Clin J Am Soc Nephrol. 2006 Sep;1(5):940-51. doi: 10.2215/CJN.00240106. Epub 2006 Jul 19. PMID 17699311